CLINICAL TRIAL: NCT05944627
Title: A Single, Dose Escalation, Optimal Dose Finding Phase I/IIa Clinical Trial to Evaluate Safety and Explore Efficacy of the Single Treatment of FURESTEM-OA Kit Inj. in Patients With Knee Osteoarthritis
Brief Title: Evaluate Safety and Explore Efficacy of FURESTEM-OA Kit Inj. in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K0701
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: FURESTEM-OA Kit Inj.; Knee Osteoarthritis Stem cell
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: Phase 1 clinical trial was an open-label. Phase 2a clinical trial was conducted in a single-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FURESTEM-OA Kit Inj. (Experimental): Subjects are slowly administered FURESTEM-OA Kit Inj. once into the knee joint cavity contained in a disposable sterile syringe mixed with Solution 1 and Solution 2 depending on the dose group assigned at the baseline (Visit 2).
  The subjects are assigned sequentially to the following 3 dose groups in Phase 1 clinical trial, and in Phase 2a clinical trial, the subjects are randomized to 1-2 dose groups below MTD determined in Phase 1.
  Interventions: Biological: FURESTEM-OA Kit Inj.
- Placebo (Placebo Comparator): Product name: Placebo of FURESTEM-OA Kit Inj. (placebo administration in Phase 2a clinical trial)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: FURESTEM-OA Kit Inj. — FURESTEM-OA Kit Inj. is a combination medical product in which FURESTEM-OA Inj. (solution 1) is the primary mode of action and CAM Inj. (solution 2) acts as an auxiliary. The product is administered after mixing solution 1 and solution 2.
  Arms: FURESTEM-OA Kit Inj.
Biological: Placebo — placebo administration in Phase 2a clinical trial
  Arms: Placebo

SUMMARY:
A Single, Dose Escalation, Optimal Dose Finding Phase I/IIa Clinical Trial to Evaluate Safety and Explore Efficacy of the Single Treatment of FURESTEM-OA Kit Inj. in Patients with Knee Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women over 19 years of age
2. Those with a body mass index (BMI) of less than 30 kg/m2 at screening
3. Those classified as ICRS grade 3 or 4 according to the International Cartilage Repair Society (ICRS) rating system through MRI examination at the time of screening
4. Those diagnosed with knee osteoarthritis according to the diagnosis criteria of the American College of Rheumatology (ACR) at the time of screening
5. Those diagnosed with Kellgren-Lawrence (K&L) grade 2-3 knee osteoarthritis (OA) at the time of screening
6. Those who do not have clinically significant abnormalities in the results of physical examination, hematologic test, blood chemistry test, or urine test
7. Those whose symptoms (pain, etc.) do not improve despite conservative therapy (drug therapy, physical therapy, etc.) for at least 12 weeks
8. Those with a 100 mm Visual Analogue Scale (VAS) score* for pain at the time of screening of 50 mm or more
9. Those who have heard and fully understood the detailed description of this clinical trial and have voluntarily decided to participate and agreed in writing to comply with the precautions

Exclusion Criteria:

1. Those who have participated in at least one other clinical trial within 4 weeks before screening and received drugs (based on the last administration date), or received medical device treatment for clinical trials
2. Those diagnosed with Kellgren-Lawrence (K&L) grade 4 knee osteoarthritis (OA) at the time of screening
3. At the time of screening, those with the results of the physical examination showing grade III (grade 0: none, grade I: 0~5 mm, grade II: 5~10 mm, grade III: >10 mm) or more ligament instability
4. Patients with osteochondritis dissecans
5. Those with hypersensitivity reactions or allergies to components of the investigational product, FURESTEM-OA Kit Inj. (combination of (FURESTEM-OA Inj.)(solution 1) + (CAM Inj.)(solution 2))
6. Those with the following confirmed medical history or surgical history / procedure history at the time of screening:

   * Patients with a history of procedure or surgery (including arthroscopy) on the target knee within 24 weeks prior to the baseline visit (Visit 2)
   * Patients who have undergone a knee joint replacement
7. Those with any of the following diseases at the time of screening:

   * Those with active infectious disease (hepatitis A/B/C (including carriers) or HIV infection that in the opinion of the investigator render those subjects as unfit to participate in this clinical trial. However, those who test positive by vaccination may participate.)
   * Those who have been determined by the investigator as having difficulty participating in this clinical trial due to a severe chronic disease (cardiovascular disease, metabolic disease, renal dysfunction, etc., excluding controlled hypertension)
   * Those with a skin disease or infection on the skin surface at the site where the investigational product is to be administered
   * Those with severe pain in other areas that may affect the determination of symptoms in the knee joint (e.g., patients with poly-articular joint pain with severe osteoarthritis symptoms in other areas (such as the hip joint))
   * Patients with other joint diseases, such as inflammatory joint diseases including rheumatoid arthritis, or infectious joint diseases such as septic arthritis, gout, recurrent pseudogout, joint fracture, acromegaly, Wilson's disease, primary osteochondrosis
   * Patients with secondary osteoarthritis due to systemic diseases such as ochronosis or hemochromatosis
   * Patients with genetic diseases such as hyperkinesia or collagen gene abnormalities
   * Patients with severe painful conditions such as Sudeck's atrophy, Paget's disease, or spinal disc herniation
8. Those with any of the following drug administration/treatment history:

   * If herbal drugs (for osteoarthritis treatment), glucosamine, chondroitin, anti-inflammatory drugs, patches, and/or other external preparations were administered within 14 days prior to the baseline visit (Visit 2) (However, participation in the clinical trial may be allowed after a sufficient wash-out period, and for glucosamine and chondroitin, participation in clinical trials is possible for health functional foods only if continuously administered from 4 weeks before screening)
   * Those who have been given drugs through intra-articular injection A. Patients who received hyaluronic acid (HA) in the target joint cavity within 12 weeks of screening B. Patients who received steroids in the target joint cavity within 12 weeks of screening C. Patients who systemically used steroids within 4 weeks of screening (except for topical application and inhalation)
   * Those who have performed physical therapy or oriental medical treatment (acupuncture, swelling, moxibustion, etc.) by a specialist for the purpose of relieving pain within 14 days prior to the baseline visit (Visit 2)
   * Those who have been given an analgesic within 14 days before administration of the investigational product, or within a time period 5 times the half-life of the analgesic.
   * Those who have been given an immunosuppressive drug (cyclosporin A or azathioprine) including antirheumatic drug (including methotrexate or antimetabolite) within 12 weeks prior to the baseline visit (Visit 2)
   * Those who have been given an anesthetic within 2 days prior to the baseline visit (Visit 2)
   * Those who have had gene therapy or cytotherapy for treatment of the knee joint
9. Those who fall under the following laboratory test results at the time of screening:

   * Serum creatinine > 2.0 mg/dL renal dysfunction
   * AST or ALT test result is more than 2.5 times the upper limit of the normal range
10. Patients with a malignant tumor (However, in the following cases, participation in the clinical trial may be allowed.)

    * Those who have been diagnosed with complete remission at least 5 years after completion of treatment for the tumor
    * If at least 1 year has elapsed since complete resection of a basal cell carcinoma/squamous cell carcinoma, radical resection of papillary thyroid cancer, or successful treatment of cervical epithelial cancer
11. Women and men of childbearing potential who are pregnant, nursing, or do not agree to perform appropriate contraception

    *Hormonal contraception (cutaneous patch, injection, oral contraceptive, etc.), intrauterine devices (loop, intrauterine system containing hormone), sterilization procedure for oneself or spouse (or partner) (vasectomy, tubal ligation, etc.), double blocking (both male (condom) and female (contraceptive diaphragm, vaginal sponge or cervical cap) must use a contraceptive device), etc.
12. Those with a history of alcohol and drug abuse within one year prior to screening
13. For other reasons, those deemed inappropriate to participate in clinical trials according to the judgment of investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-07-06 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of FURESTEM-OA Kit Inj. | 4 weeks follow-up after treatment
  Maximum Tolerated Dose (MTD) identification based on Dose Limiting Toxicities (DLTs) evaluation Evaluation of adverse events

SECONDARY OUTCOMES:
Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS) score | week 1, week 4, week 8, week 12, week 16, week 20 and week 24 after treatment
Rate and amount of changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | week 1, week 4, week 8, week 12, week 16, week 20 and week 24 after treatment
Changes in 100 mm VAS score | week 1, week 4, week 8, week 12, week 16, week 20 and week 24 after treatment
Changes in the International Knee Documentation Committee Scoring System (IKDC) score | week 1, week 4, week 8, week 12, week 16, week 20 and week 24 after treatment
Evaluation of K&L grade | week 24 after treatment
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score | week 24 after treatment
Whole-Organ Magnetic Resonance Imaging Score (WORMS) score | week 24 after treatment
Rate and amount of changes in biomarker values | week 1, week 4, week 8, week 12, week 16, week 20 and week 24 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Ho Yoon, professor (CI), Principal Investigator — Kyung Hee University Hospital; Sang Hak Lee, professor, Principal Investigator — Gangdong Kyunghee University Hospital